CLINICAL TRIAL: NCT04270227
Title: Does Physical Activity Level Depend on Exercise Perception and Body Awareness
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal investigator, Istanbul Medipol University Hospital
Other Study IDs: Body awareness_Exercise
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Healthy
MeSH Terms: interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey study — The questionnaire including Exercise Benefits / Barriers Scale, IPAQ (International Physical Activity Survey), The Bady Awareness questionnaire and demographic information will be filled in one time by face-to-face interview method.

SUMMARY:
Healthy volunteers between the ages of 18-25 who will not have any problems preventing physical activity will be included among the university students. The criteria for not being included in the study were determined as being diagnosed with any disease that impedes physical activity and not wanting to participate in the study. Participation in the investigator's study is completely voluntary. Individuals who do not wish to participate in the study will be excluded. Cases with missing survey and demographic information will be excluded from the study. The planned study is a cross-sectional study.

ELIGIBILITY:
Inclusion Criteria:

* Not having any problems preventing physical activity
* No identified chronic disease
* Being between the ages of 18-25

Exclusion Criteria:

-Not want to participate in the study

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: Young healthy adults
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Body awareness scale (Body awareness questionnaire-Turkish) | 15 minutes
  It is a questionnaire consisting of four subgroups (changes in the body process, sleep-wake cycle, prediction at the onset of the disease, prediction of body responses) and a total of 18 expressions aimed at determining the normal or abnormal sensitivity level of the body composition. The participant is asked to score between one and seven numbers for each statement. In the survey, the ratings are made as total points. The high score shows that body sensitivity is better.

SECONDARY OUTCOMES:
Exercise Benefits/Barriers Scale | 15 minutes
  It is a 43-item questionnaire using the 4-item Likert scale. The score varies between 43 and 172. High scores on the benefits scale show the perceived benefits of physical activity, while high scores on the barrier scale show that perceived barriers to physical activity are low.
International Physical Activity Questionnaire Short Form | 15 minutes
  Physical activity levels of the participants according to the total physical activity score; It was classified as physically inactive (3000MET-min / hf) and low physical activity level (600-3000 MET-min / hf) with sufficient physical activity level (> 3000MET-min / hf).

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Pehli̇van, Istanbul, Üsküdar, Turkey (Türkiye)